CLINICAL TRIAL: NCT02964390
Title: Assessment of Safety and Efficacy of Balloon Pulmonary Angioplasty in Non-operable CTEPH Patients
Brief Title: Balloon Pulmonary Angioplasty in Non-operable CTEPH Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Department of Pulmonary Circulation and Thromboembolic Diseases, Medical Center for Postgraduate Med (Other)
Responsible Party: Principal Investigator, Marcin Kurzyna, MD, PhD, Department of Pulmonary Circulation and Thromboembolic Diseases, Medical Center for Postgraduate Med
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 002
Record Dates: First submitted 2016-09-06; First posted 2016-11-16 (Estimated); Last update posted 2021-08-19 (Actual); Status verified 2021-08

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension
Keywords: CTEPH; balloon pulmonary angioplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Balloon Pulmonary Angioplasty (Experimental): This arm includes patients qualified to BPA procedure. They have a baseline workup performed before the initiation of BPA treatment and had a follow up examination from 3 to 6 months after the last BPA session.
  Interventions: Procedure: Balloon Pulmonary Angioplasty

INTERVENTIONS:
Procedure: Balloon Pulmonary Angioplasty
  Other Names: BPA

SUMMARY:
Balloon pulmonary angioplasty (BPA) emerged as a potential therapeutic option for non-operable patients with chronic thromboembolic pulmonary hypertension (CTEPH).

The aim of this study was to evaluate the safety and efficacy of BPA in patients disqualified from surgery or suffered from persistent CTEPH despite pulmonary endarterectomy.

This is a interventional study analyzing the benefits and the risk of BPA. Clinical evaluation, including: functional capacity, 6-minutes walking test, haemodynamics, biomarkers, cardiopulmonary exercise test, echocardiography, electrocardiography and QoL assessment with Short Form 36 (SF36) questionnaire was performed before the initiation therapy of BPA, and 3-6 months after last session of BPA.

DETAILED DESCRIPTION:
Chronic thromboembolic pulmonary hypertension (CTEPH) is a rare but potentially life-threatening disease of the pulmonary circulation. Management of CTEPH requires precise differential diagnosis, long life anticoagulation when confirmed and qualification for surgical treatment by an experienced multidisciplinary team. The gold standard of treatment in operable patients is pulmonary endarterectomy (PEA), which is highly effective in restoring functional status and improving life expectancy. Nevertheless, even in the leading CTEPH referral centres almost 50% patients remain on medical treatment alone, with grim perspectives regarding life quality and expectancy. Recently, balloon pulmonary angioplasty (BPA) has emerged as a promising new interventional option in non-operable CTEPH.

The development BPA was far from rapid. It took 13 years from the first case-report to the publication of a first series of 17 patients treated with BPA in Boston/US and another 13 years until the results of first European series of 20 patients has been reported from Oslo/Norway. In Poland BPA was started to perform in non-operable CTEPH patients in 2013, motivated by their expected poor prognosis, when compared to those to whom surgical PEA was offered.

The aim of this study is an analysis of efficacy and safety of BPA procedure.

The BPA is performed by two senior interventional specialist - cardiologist and radiologist with extensive experience in coronary, pulmonary and general vessel interventions supported by perfusion nurse. All patients undergoing BPA are given informed consent before the first BPA intervention. The limited experience with and experimental nature of BPA are emphasised to candidates.

A standard BPA procedure is typically performed from the right femoral vein, with anticoagulation of unfractionated heparin in periprocedural period. A long (70 or 90 cm) sheath is introduced into the pulmonary trunk with support of pigtail catheter. Selective and super-selective catheterisation of lobar arteries, segmental and when appropriate subsegmental arteries is performed to demonstrate variety of clots: "webs", "rings", "occlusions", "pouch" lesions and reduction of parenchymal opacification after injection of vascular contrast medium. Balloon catheters (diameter 1.25-6.0 mm) are positioned over the selected lesion and dilated for several seconds. Immediate selective angiography is performed after dilation to confirm satisfactory results which presented the improvement of contrast medium distribution and venous return. Control angiography is done to rule out residual stenosis or signs of vessel injury. Following BPA procedure, patients are moved to ICU for 48 h surveillance.

Right before the initiation of BPA and during 3-6 months after last session, a full workup is made, including: World Health Organization (WHO) functional class, 6-minute walking test (6MWT), concentration of biomarkers (NT-proBNP, Troponin T, sST2), cardiopulmonary exercise test, echocardiography, electrocardiography and right heart catheterization including measurements of right atrial pressure (RAP), pulmonary artery pressure (PAP), pulmonary capillary wedge pressure (PCWP), cardiac output (CO), cardiac index (CI), pulmonary vascular resistance (PVR), mixed venous oxygenation (MVsat.O2) and systemic oxygenation (AOsatO2). Additionally patients fill in the Short Form 36 (SF36) quality of life questionnaire before initiation of BPA and 3-6 months after last session.

ELIGIBILITY:
Inclusion Criteria:

* diagnosed with CTEPH according to ESC Guidelines
* WHO functional capacity ≥ II
* documented period of anticoagulation > 6 months after the episode of Pulmonary Embolism,

Exclusion Criteria:

* age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-07; Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety of BPA procedure. | From initiation of BPA to 3-6 months after last session
  Surveillance of complications including: vessel injury, desaturation, cough, mild hemoptysis (<50ml), severe hemoptysis (>50ml), reperfusion pulmonary injury, death.
Improvement of haemodynamics caused by series of BPA. | From initiation of BPA to 3-6 months after last session
  Measurements taken during right heart catheterization in at least 25 patients with accomplished interventional treatment of BPA. The measurements will include pulmonary artery pressure - PAP [mmHg].
Improvement of functional capacity caused by series of BPA. | From initiation of BPA to 3-6 months after last session.
  Examined using World Health Organization (WHO) functional capacity classification is evaluated by physician in every patient, on admission and follow up.
Improvement of NT-proBNP caused by series of BPA. | From initiation of BPA to 3-6 months after last session.
  Baseline measurements of the concentration of NT-proBNP [pg/ml] in at least 25 subjects who accomplished their invasive treatment.
Improvement of six minutes walk test caused by series of BPA. | From initiation of BPA to 3-6 months after last session.
  Six minutes walking test - 6MWT is performed according to European Society of Cardiology (ESC) guidelines. The baseline distance [meters] covered during the 6MWT will be compared to the follow up value in patients (at least 25) who accomplished their invasive treatment of BPA.

CONTACTS AND LOCATIONS:
Overall Officials: Marcin Kurzyna, MD,PhD, Principal Investigator — European Health Center Otwock
Locations (1):
- European Health Center Otwock, Otwock, Poland

IPD SHARING:
Plan to Share IPD: No